CLINICAL TRIAL: NCT07256938
Title: Effect of Clonidine Additive to suprascapular_ Costoclavicular Versus Standard Interscalene Block in Arthroscopic Shoulder Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Fathy Khedr, residant doctor at Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: clonidine + suprascapular
Record Dates: First submitted 2025-11-21; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Arthroscopic Shoulder Surgeries
MeSH Terms: interventions — Bupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): US-guided costoclavicular block
  Interventions: Drug: Bupivacaine 0.5% (hyperbaric); Procedure: US-guided costoclavicular block; Procedure: Interscalene brachial plexus block; Drug: clonidine 1 mg / kg
- Group B (Active Comparator): US-guided interscalene brachial plexus block
  Interventions: Drug: Bupivacaine 0.5% (hyperbaric); Procedure: US-guided costoclavicular block; Drug: clonidine 1 mg / kg; Procedure: single shot US-guided suprascapular nerve block

INTERVENTIONS:
Drug: Bupivacaine 0.5% (hyperbaric) — 5 mL bupivacaine 0.5%,
Procedure: US-guided costoclavicular block — US-guided costoclavicular block
Procedure: Interscalene brachial plexus block — single shot US-guided interscalene brachial plexus block
  Arms: Group A
Drug: clonidine 1 mg / kg — clonidine 1 mg / kg
Procedure: single shot US-guided suprascapular nerve block — single shot US-guided suprascapular nerve block
  Arms: Group B

SUMMARY:
Postoperative analgesia for shoulder surgery is typically achieved by providing an interscalene brachial plexus block. However, a very common side effect of this block is hemi-diaphragmatic paralysis, a state which may not be tolerated in patients with pulmonary conditions such as COPD.

Recently, clinicians have explored new ways to provide satisfactory analgesia while minimizing the pulmonary side effects of the interscalene nerve block. One of these solutions might be to offer the patient a suprascapular nerve block combined to costoclavicular block. Since these blocks are performed lower in the neck or under the clavicle, the phrenic nerve is less likely to be blocked. Thus, fewer respiratory side effects have been reported when using such blocks.

Hypothesis The main hypothesis of this study is that the addition of clonidine to suprascapular block combined with costoclavicular block is not inferior to the standard interscalene brachial plexus block in terms of postoperative analgesia. We postulate that pain score postoperatively and opioid requirements will not differ significantly in patients who receive either block.

Our secondary objectives will consist in looking at the differences in intraoperative , arm motor block , diaphragmatic paresis , patient satisfaction and time for readiness to discharge from PACU .we hypothesize that these outcomes will be similar in both groups , with the exception of a potential reduction in arm motor block and diaphragmatic paresis in the combined suprascapular and costoclavicular block group The primary objective of this study will be to evaluate the postoperative pain score during arthroscopic shoulder surgery assessed by the pain score when comparing the effect of addition of clonidine to suprascapular_costoclavicular versus standard interscalene

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1,2,3. Age( 18-60) years Elective shoulder arthroscopic surgery under general anesthesia and nerve bloc performed preoperatively

Exclusion Criteria:

* Patient refusal Coagulation disorders. Anatomical disorders and/or neuropathic disease. BMI above 40. History of substance abuse. Chronic use of psychotropic and/or opioid. History of psychiatric diseases needing treatment. Contraindications to nerve block for shoulder surgery. Allergy to fentanil or any drug in the study protocol. Failure of nerve block performed in the preoperative block room when tested prior to entering the operating room (i.e. lack of loss of sensation to ice at the shoulder incision level).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | 24 hours postoperative
  to evaluate postoperative pain score during arthroscopic shoulder surgery assessed by the pain score when comparing the combined suprascapular and costoclavicular nerve blocks to the interscalene brachial plexus block